CLINICAL TRIAL: NCT02740920
Title: A Phase II Study of the Assessment of Response to Pembrolizumab in Metastatic Melanoma: CT Texture Analysis as a Predictive Biomarker
Brief Title: Response to Pembrolizumab in Metastatic Melanoma: Computed Tomography Texture Analysis as a Predictive Biomarker
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I225
Record Dates: First submitted 2016-04-06; First posted 2016-04-15 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): 200mg IV Day 1 every 3 weeks.
  Interventions: Drug: Pembrolizumab; Procedure: CT Scan

INTERVENTIONS:
Drug: Pembrolizumab
Procedure: CT Scan

SUMMARY:
Studies have shown that the study drug, pembrolizumab, works by helping the immune system. In this way, pembrolizumab may help to slow the growth of melanoma or may cause cancer cells to die. Compared to standard treatments, pembrolizumab seems to lengthen the time patients lived overall and the time without their cancer getting worse.

DETAILED DESCRIPTION:
The main purpose of this study is to find out if a type of CT (computed topography) scan can help to know if pembrolizumab is working. This CT scan (called Texture Analysis) looks at the tumour in fine detail. The use of this type of CT scan has not been studied in patients with metastatic melanoma. Investigators want to see if this CT scan will show if some patients being treated with pembrolizumab respond better than others.

One of the other purposes is to compare the costs within this trial to costs of the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma that is recurrent/metastatic and not amenable to potentially curative surgery.
* Presence of clinically and/or radiologically documented disease based on RECIST 1.1. At least one site of disease must be unidimensionally measurable by contrast-enhanced CT scan as follows:

CT scan (with slice thickness of ≤ 5 mm) ≥ 10 mm --> longest diameter Lymph nodes by CT scan ≥ 15 mm --> measured in short axis

* Age ≥ 18 years.
* ECOG Performance Status of 0 to 1.
* Previous Therapy

Surgery:

Previous surgery is permitted provided that it has been at least 21 days prior to patient registration and that wound healing has occurred.

Systemic Therapy:

Patients may not have received any prior systemic therapy for metastatic melanoma.

Radiation:

Palliative radiation is permitted provided > 7 days has elapsed between last dose and enrollment on the trial.

* Laboratory Requirements Absolute neutrophils ≥ 1.5 x 10^9/L Platelets ≥ 100 x 10^9/L Hemoglobin ≥ 90 g/L or ≥ 5.6 mmol/L (without transfusion or EPO dependency) Serum creatinine or measured or calculated creatinine: ≤1.5 x ULN or ≥ 60 mL/min for subject with creatinine clearance levels > 1.5 x ULN Serum Total Bilirubin ≤ 1.5 x ULN or Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 x ULN AST and ALT ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver mets) Albumin ≥ 25 g/L
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method.
* Women of childbearing potential will have a serum or urine pregnancy test within 7 days prior to registration to determine eligibility.
* Patient consent must be obtained according to local Institutional and/or University Human Experimental Committee requirements.
* Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating centre.

Exclusion Criteria:

* Patients who have received prior systemic treatment for metastatic melanoma.
* Patients with known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Patients with a known history of or known positive for Hepatitis B (HBsAg reactive) or Hepatitis C (HCV RNA [qualitative] is detected). Patients with unknown history of Hepatitis B virus (HBV) or Hepatitis C virus (HCV) will require screening.
* Patients with previously treated brain metastases may participate provided they are stable with no evidence of enlargement following radiation treatment and no acute radiation toxicity OR no evidence of enlargement at least 4 weeks prior to the first dose of study drug if untreated and are off systemic steroids for at least two weeks.
* Patients who are pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the pre-screening or screening visit through 4 months after the last dose of trial treatment.
* Patients who previously had a severe hypersensitivity reaction to treatment with another mAb.
* Patients with an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. (Only patients on active treatment are ineligible).
* Patients with a history of a malignancy (other than the disease under treatment in the study) within 5 years prior to first study drug administration.
* Patients on any systemic corticosteroid therapy within one week before the planned date for first dose of treatment or on any other form of immunosuppressive medication.
* Patients with an allergy to iodinated contrast media used for CT.
* Patients with a known history of active TB (Bacillus Tuberculosis).
* Patients with evidence of interstitial lung disease;
* Patients with known history of, or any evidence of active, non-infectious pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Petrella, Study Chair — Sunnybrook Health Sciences Centre, Toronto ON
Locations (5):
- Canada (5):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab: 200mg IV Day 1 every 3 weeks.
  Pembrolizumab
  CT Scan
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled into the study
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 65 [37 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 2
Performance status [Count of Participants; unit: Participants] — Measure Description: The scale was developed by the Eastern Cooperative Oncology Group (ECOG) Grade 0: Fully active, able to carry on all pre-disease performance without restriction Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    Grade 0 | 6
    Grade 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Tumor Texture by CT Scan
Description: To assess whether tumour texture parameters from a CT scan can differentiate patients who do and who do not respond to treatment with pembrolizumab. Trial closed due to slow accrual, analysis was no done for the primary outcome because data were not collected.
Time Frame: 12 months
Population: Trial closed due to slow accrual, analysis was no done for the primary outcome because data were not collected.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Response Rate Assessed by CT Scan
Description: To determine the overall response rate (complete + partial response)/total number of patients.
  Response and progression will be evaluated in this study using the revised international criteria (1.1) proposed by the RECIST (Response Evaluation Criteria in Solid Tumours) committee as well as the modified iRECIST guidelines. Response were assessed by CT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 24 months
Population: All patients who received the protocol treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 9
Participants
  Number of Response | 2
  Nomuber of non-response | 7

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 5/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=9)
Fever (General disorders) | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1
Other neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Other nervous system disorders (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=9)
Chest pain - cardiac (Cardiac disorders) | 1
Blurred vision (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Other gastrointestinal disorders (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 4
Fever (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 2
Other infections and infestations (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 3
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Other neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Other nervous system disorders (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT02740920/Prot_SAP_000.pdf